CLINICAL TRIAL: NCT05666271
Title: Radiofrequency Ablation for Small Hepatocellular Carcinoma Using Octopus MP Electrodes or Octopus Electrodes With Adjustable Tips: A Prospective Observational Study
Brief Title: Radiofrequency Ablation for Hepatocellular Carcinoma Using Octopus MP Electrodes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: 2208-116-1351
Record Dates: First submitted 2022-12-18; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation will be performed by using the Octopus MP electrodes. It is a method of directly measuring the temperature near the surrounding tissue of the target tumor using the Octopus MP electrode, and stopping ablation when the temperature rises above 60 degrees to prevent adjacent organ (gallbladder, gastrointestinal tracts, diaphragm, and heart). If the shape of the tumor is elliptical or irregular rather than circular, using an adjustable tip that can change the length of the active tip of the electrode according to the size of the tumor has the advantage of tailoring the ablation zone.

SUMMARY:
This study is to investigate the therapeutic effect and treatment results of radiofrequency ablation using the Octopus MP electrode capable of temperature monitoring and drug injection and a variable-length electrode for treatment of small hepatocellular carcinomas (≤ 3cm).

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class A or B
* chronic hepatitis B or chronic hepatitis C or liver cirrhosis
* presence of hepatocellular carcinoma (HCC) after confirmed by pathology or imaging studies including contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) according to the Korean Liver Cancer Study Group (KLCSG)-National Cancer Center (NCC) Korea practice guidelines.
* up to 3 lesions, each greater than less than or equal to 3 cm at the time of locoregional treatment.

Exclusion Criteria:

* number of recurrent HCCs, more than 3
* largest HCC size over 3 cm
* presence of vascular invasion by HCC
* platelet count less than 40,000 per mm3 or International Normalized Ratio (INR) prolongation over 50%
* presence of extrahepatic metastasis

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred for radiofrequency ablation for the treatment of small hepatocellular carcinomas (equal or less than 3 cm) located in the periphery of the liver (within 5 cm from the liver capsule) on preprocedural computed tomography or magnetic resonance imaging.
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Adjacent organ thermal injury rate | Immediately after radiofrequency ablation
  Evaluate adjacent organ thermal injury rate by immediate follow-up computed tomography after radiofrequency ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No